CLINICAL TRIAL: NCT01134172
Title: Breast Cancer and the Workforce: Ethnic Differences in the Impact of Breast Cancer on Employment Status, Financial Situation, and Quality of Life (BCW)
Brief Title: Ethnic Differences in the Impact of Breast Cancer on Employment Status, Financial Situation, and Quality of Life
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: The City College of New York (Other); NYC Health & Hospitals/ Lincoln Medical Center (Unknown); New York Presbyterian Queens (Unknown); New York City Health and Hospitals Corporation (Other); Queens Medical Associates (Unknown)
Responsible Party: Sponsor
Other Study IDs: 10-071
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Sociodemographic; Ethnicity; Work-related; Health system; QOL; Questionnaires; 10-071
MeSH Terms: conditions — Breast Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Breast cancer survivors: Women being treated for stage I-III breast cancer who were employed prior to this diagnosis will be recruited in their physicians' offices.
  Interventions: Behavioral: survey web-based or telephone interview
- Comparison group: Peer controls will be nominated by participants in the breast cancer survivor group or recruited by community outreach and matched for age, language, and ethnicity. This cohort is no longer recruiting.
  Interventions: Behavioral: survey web-based or telephone interview

INTERVENTIONS:
Behavioral: survey web-based or telephone interview — Patients will be asked to complete a questionnaire at baseline, and then one at follow up, 3-4 months after treatment completion. The patient will be contacted one and two years after the completion of their follow up questionnaire for a brief one-question survey regarding current employment status. A member of the study team will call a subset of patients who have completed both baseline and follow-up surveys to clarify responses to previous questions. Patients will be considered lost to follow- up if surveys A or C have not been completed two years from the participant's consent date (participants who enroll but do not complete survey A are not prompted for survey C). Deviations will not be filed until the end of the study, as there are opportunities over the course of study follow- up to collect previously missing information.
  Groups: Breast cancer survivors
Behavioral: survey web-based or telephone interview — Patients will be asked to complete a questionnaire at baseline, and then one at follow up, 3-4 months after treatment completion. All three follow-up contact methods (email, postcard, call) contain the same question regarding current employment status with minor modifications in formatting. However, the employment question asked in all three follow-up contact methods is shown in the Postcard_Template document. Due to the recent COVID-19 pandemic study staff will be working from home. Therefore, calls will be made via MSK-approved platforms (e.g. Jabber, etc.). Participants who express concerns or request assistance related to COVID-19 will be referred to publicly available resources as needed (e.g., call 311 for access to health care or food panties, etc.) and will be noted in internal tracking logs. The data collected for these internal tracking logs will be managed through a REDCap database.
  Groups: Comparison group

SUMMARY:
The purpose of this study is to learn more about how being treated for breast cancer affects patients' employment, financial situation, and quality of life on a short-term basis and on a long term basis. Most studies of employment after breast cancer have focused on Caucasian women.This study will evaluate the impact of breast cancer on the lives of women from different ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

Breast cancer survivors

* Pathologic diagnosis of stage I-III breast cancer
* Paid employment (full time or part time) at time of consent or in the three months prior to diagnosis
* Age 18 to 64 years (inclusive)
* The ability to give informed consent in Chinese (Mandarin), English, Korean, or Spanish.at MSK, New York Presbyterian Queens and Queens Medical Associates At NYC Health & Hospitals/ Lincoln Medical Center, patients must be able to give consent in English or Spanish.
* At the time of enrollment, participants must still be undergoing chemotherapy, undergoing radiation therapy, or planning surgery unless surgery is to be the only treatment modality. Those for whom treatment consists of surgery alone may have had their operation no more than 2 months prior to study enrollment. Participants need not have undergone surgical reconstruction prior to enrollment if the plan is to delay this procedure until after primary treatment is completed.

Comparison group

Paid employment (full time or part time) at the time of consent

* Age 18 to 64 years (inclusive) and within an age range that is 5 years above or below that of the nominating or matched survivor
* The ability to give informed consent in the same language as the nominating survivor
* Membership in the same ethnic group as the nominating survivor
* Not treated for cancer in the past year (other than non-melanoma skin cancer)

Exclusion Criteria:

* N/A

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will recruit participants from Memorial Sloan-Kettering Cancer Center (MSKCC), four of its community-based outpatient treatment centers, and four urban community hospitals and clinics that serve large populations of ethnic minorities in New York City. The MSKCC outpatient regional sites are located in New Jersey (Basking Ridge, Monmouth) and New York, with two in Long Island (Commack and Rockville Centre) and another in Westchester County.
Sampling Method: Non-Probability Sample
Enrollment: 935 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
To compare the impact of breast cancer on (a) employment status, (b) financial situation, and (c) QoL. | 3 years

SECONDARY OUTCOMES:
To identify barriers to employment and correlates of employment status, financial situation, and QoL. | 3 years
To develop the methodology to evaluate discrimination in the labor market using a validated instrument and to determine whether or not labor market discrimination is exacerbated by a diagnosis of breast cancer. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Blinder, M.D., M.Sc., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (12):
- United States (12):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Woodhull Medical and Mental Health Center, Brooklyn, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Queens Medical Associates, Fresh Meadows, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering at Ralph Lauren, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Bellevue Hospital Center, New York, New York
  - New York Presbyterian Queens, Queens, New York
  - NYC Health & Hospitals /Lincoln Medical Center, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm